CLINICAL TRIAL: NCT06412172
Title: The Natural History and Biological Study of Pulmonary Recurrent Respiratory Papillomatosis (pRRP)
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara Pai, MD, PhD, Associate Surgeon, Massachusetts General Hospital
Other Study IDs: HIC# 2000037079
Record Dates: First submitted 2024-04-14; First posted 2024-05-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Respiratory Papillomatosis; Pulmonary Neoplasm
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin embedded tissue and/or unstained slides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recurrent respiratory papillomatosis (RRP) is an orphan disease that affects approximately 20,000 people in the United States and is caused by infection with human papillomavirus (HPV) types 6 and 11. Since RRP is an orphan disease, it is an understudied disease entity with correspondingly few treatment options. The investigators hypothesize that by understanding the biology of RRP and the failed host immune responses against HPV, novel and rational therapies can be developed. This study will examine the genetic and immunologic alterations found in these rare tumors and distant metastatic involved sites (such as the lung) in patients diagnosed with RRP.

DETAILED DESCRIPTION:
Since RRP is an orphan disease, any single institution or hospital treats a limited number of RRP patients. The primary purpose for establishing a tissue repository is to collect RRP tissue from various institutions and hospitals and to provide investigators access to a large number of RRP tissues to perform genetic and immunologic studies of these rare tumors. This is both a prospective and retrospective tissue collection repository. Tissue that will be collected will include excess fresh or archived human tissue, either normal or pathological, that was removed as part of standard of care clinical procedures and/or during procedures performed for separate research purposes, such as a therapeutic clinical trial. Prospectively collected and archived pathology samples will be obtained under informed consent from those patients who are still living. The tissue repository will be de-identified. The PI and the RRP Foundation will collaborate and serve as the gatekeepers of the repository and oversee any tissue requests. Any academic collaborator(s) or for-profit collaborator(s) can request access to the tissue specimens. The investigator or collaborators should submit a letter to express interest in obtaining tissue from the tissue repository to the RRP Foundation and the PI.

ELIGIBILITY:
Inclusion Criteria:

* History of HPV-associated Recurrent Respiratory Papillomatosis
* Has pulmonary lesions

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HPV-associated RRP. The investigators will collect, store, and study primary tissue and distant anatomic sites of disease which were removed as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2030-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with HPV 6 or 11 infection in the pulmonary lesions | 24 months
  HPV 6 and 11 genotyping will be done via polymerase chain reaction
Number of Participants with different mutational profiles in the matched laryngeal and pulmonary lesions | 24 months
  Sequencing of the HPV genome in the matched laryngeal and pulmonary lesions will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pai, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States